CLINICAL TRIAL: NCT00719004
Title: Sonographic Features of Normal Soft Tissues of the Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gandikota Girish, MD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00007286
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Foot Disease; Healthy
Keywords: Anatomy; Foot; Sonography; Medical
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normals (Experimental): Normal volunteers having Ultrasound scan of foot.
  Interventions: Procedure: Ultrasound of the foot

INTERVENTIONS:
Procedure: Ultrasound of the foot — These volunteers will have one ultrasound scan of each foot

SUMMARY:
The purpose of this study is to study normal sonographic(ultrasound)anatomy of the soft tissues of the foot in normal volunteers.

DETAILED DESCRIPTION:
To study normal sonographic anatomy of soft tissues of the foot [which include Extensor retinaculum, sinus tarsi, ligaments and tendons, spring ligament and their attachments to underlying bones] in asymptomatic individuals/volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* no disease or abnormality of the feet

Exclusion Criteria:

* abnormality of the feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Clinical relevance of understanding the anatomy will help in early and accurate identification of pathology. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gandikota Girish, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No